CLINICAL TRIAL: NCT04800588
Title: Computerized Tests of Cognitive Decline in Presymptomatic Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurobehavioral Systems, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4R44AG062076 (NIH)
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Cognitive Decline; Aging
Keywords: Aging; Elderly; Alzheimer's disease; Cognition; Computerized; Testing
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Older participant group (Experimental): We will evaluate the performance of healthy older participants (N = 300, age range 60 to 89 years) for three days at enrollment and then at 6-month intervals for three years thereafter. The goal is to characterize changes in performance to aging and task experience in a group of older subjects.
  Interventions: Diagnostic Test: California Cognitive Assessment Battery
- CCAB vs. manual test group (Experimental): We will compare the performance of normal participants (N = 100, age range 18 to 89) on computerized and manually administered cognitive tasks.
  Interventions: Diagnostic Test: California Cognitive Assessment Battery
- Test-Retest Reliability group (Experimental): We will gather normative data from participants across the age range (N = 100, ages 18 to 89) for three days at enrollment, to better characterize test-retest reliability scores on Day 1 tasks.
  Interventions: Diagnostic Test: California Cognitive Assessment Battery
- Health Disparities group (Experimental): We will evaluate the performance of healthy older participants (N = 1200, age range 50 to 89 years) for three days at enrollment and then at 6-month intervals for three years thereafter. In the aim of better understanding health disparities in cognitive testing, this group will be divided into four cohorts: 300 African American participants; 300 Asian American participants; 300 Latino English-speaking participants; and 300 Latino Spanish-speaking participants, who will complete a Spanish translation of our computerized cognitive tests.
  Interventions: Diagnostic Test: California Cognitive Assessment Battery

INTERVENTIONS:
Diagnostic Test: California Cognitive Assessment Battery — The California Cognitive Assessment Battery (CCAB) is a collection of computerized cognitive tests that will be telemedically administered to participants in their homes using a tablet computer and accessories provided by the research team. Testing may also occur in research laboratories. Previous versions of CCAB tests have been described in 16 manuscripts which describe (a) the psychometric characteristics of normative data collected in large participant populations (300 to 2,300 subjects for different tests) and (b) the sensitivity of CCAB tests for detecting performance abnormalities in patients with traumatic brain injury (TBI) and in control participants simulating the cognitive deficits that follow mild TBI.
  Other Names: CCAB

SUMMARY:
The investigators will study performance on computerized cognitive tasks in healthy participants of different ages to gather normative data for newly developed computerized cognitive tests. These tests are designed to permit the early detection of individuals at risk of age-related cognitive decline.

DETAILED DESCRIPTION:
In Group A, the investigators will evaluate the performance of healthy older participants (N = 300, age range 60 to 89 years) for three days at enrollment and then at 6-month intervals for three years thereafter. The goal is to characterize changes in performance to aging and task experience in a group of older subjects.

In Group B, the investigators will compare the performance of normal participants (N = 100, age range 18 to 89) on computerized and manually administered cognitive tasks.

In Group C, the investigators will gather normative data from participants across the age range (N = 100, ages 18 to 89) for three days at enrollment, to better characterize test-retest reliability scores on Day 1 tasks.

In Group D, the investigators will evaluate the performance of healthy older participants (N = 1200, age range 60 to 89 years) for three days at enrollment and then at 6-month intervals for three years thereafter. In the aim of better understanding health disparities in cognitive testing, this group will be divided into four cohorts: 300 African American participants; 300 Asian American participants; 300 Latino English-speaking participants; and 300 Latino Spanish-speaking participants, who will complete a Spanish translation of our computerized cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to use computer mouse and touch screen
* Must speak English as a primary language
* Must speak Spanish as a primary language (for Latino participants completing our Spanish translation)

Exclusion Criteria:

* History of psychiatric disorder
* History of stroke or transient ischemic attack
* History of substance abuse
* History of medical or sensory disorders that are incompatible with effective testing
* History of traumatic brain injury with hospitalization and extended loss of consciousness
* History of epilepsy
* History of depression or anxiety

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal normative data collection from healthy participants | Longitudinal testing at six-month intervals
  Multiple behavioral outcome measures will be obtained from each cognitive test including measures of response time (in milliseconds) and accuracy (in percent correct). Recordings of subject's verbal responses will also be analyzed phonologically and automatically transcribed to permit the lexical, syntactic, and semantic analysis of speech output. Questionnaire data will be used to identify factors that may influence performance on the cognitive tests. The primary outcome measures are the scores obtained during enrollment testing that predict a decline in longitudinal performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurobehavioral Systems, Inc., Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woods DL, Kishiyamaa MM, Lund EW, Herron TJ, Edwards B, Poliva O, Hink RF, Reed B. Improving digit span assessment of short-term verbal memory. J Clin Exp Neuropsychol. 2011 Jan;33(1):101-11. doi: 10.1080/13803395.2010.493149. PMID 20680884
- [Background] Woods DL, Herron TJ, Yund EW, Hink RF, Kishiyama MM, Reed B. Computerized analysis of error patterns in digit span recall. J Clin Exp Neuropsychol. 2011 Aug;33(7):721-34. doi: 10.1080/13803395.2010.550602. PMID 21957866
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. The Effects of Repeat Testing, Malingering, and Traumatic Brain Injury on Computerized Measures of Visuospatial Memory Span. Front Hum Neurosci. 2016 Jan 5;9:690. doi: 10.3389/fnhum.2015.00690. eCollection 2015. PMID 26779001
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. An improved spatial span test of visuospatial memory. Memory. 2016 Sep;24(8):1142-55. doi: 10.1080/09658211.2015.1076849. Epub 2015 Sep 11. PMID 26357906
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. The Bay Area Verbal Learning Test (BAVLT): Normative Data and the Effects of Repeated Testing, Simulated Malingering, and Traumatic Brain Injury. Front Hum Neurosci. 2017 Jan 12;10:654. doi: 10.3389/fnhum.2016.00654. eCollection 2016. PMID 28127280
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW, Reed B. The Dyad-Adaptive Paced Auditory Serial Addition Test (DA-PASAT): Normative data and the effects of repeated testing, simulated malingering, and traumatic brain injury. PLoS One. 2018 Apr 20;13(4):e0178148. doi: 10.1371/journal.pone.0178148. eCollection 2018. PMID 29677192
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. The Effects of Aging, Malingering, and Traumatic Brain Injury on Computerized Trail-Making Test Performance. PLoS One. 2015 Jun 10;10(6):e0124345. doi: 10.1371/journal.pone.0124345. eCollection 2015. PMID 26060999
- [Background] Woods DL, Wyma JM, Yund EW, Herron TJ, Reed B. Factors influencing the latency of simple reaction time. Front Hum Neurosci. 2015 Mar 26;9:131. doi: 10.3389/fnhum.2015.00131. eCollection 2015. PMID 25859198
- [Background] Woods DL, Wyma JM, Yund EW, Herron TJ. The Effects of Repeated Testing, Simulated Malingering, and Traumatic Brain Injury on High-Precision Measures of Simple Visual Reaction Time. Front Hum Neurosci. 2015 Nov 9;9:540. doi: 10.3389/fnhum.2015.00540. eCollection 2015. PMID 26617505
- [Background] Hubel KA, Reed B, Yund EW, Herron TJ, Woods DL. Computerized measures of finger tapping: effects of hand dominance, age, and sex. Percept Mot Skills. 2013 Jun;116(3):929-52. doi: 10.2466/25.29.PMS.116.3.929-952. PMID 24175464
- [Background] Hubel KA, Yund EW, Herron TJ, Woods DL. Computerized measures of finger tapping: reliability, malingering and traumatic brain injury. J Clin Exp Neuropsychol. 2013;35(7):745-58. doi: 10.1080/13803395.2013.824070. Epub 2013 Aug 15. PMID 23947782
- [Background] Woods DL, Wyma JM, Yund EW, Herron TJ. The Effects of Repeated Testing, Simulated Malingering, and Traumatic Brain Injury on Visual Choice Reaction Time. Front Hum Neurosci. 2015 Nov 24;9:595. doi: 10.3389/fnhum.2015.00595. eCollection 2015. PMID 26635569
- [Background] Woods DL, Wyma JM, Yund EW, Herron TJ, Reed B. Age-related slowing of response selection and production in a visual choice reaction time task. Front Hum Neurosci. 2015 Apr 23;9:193. doi: 10.3389/fnhum.2015.00193. eCollection 2015. PMID 25954175
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. Computerized Analysis of Verbal Fluency: Normative Data and the Effects of Repeated Testing, Simulated Malingering, and Traumatic Brain Injury. PLoS One. 2016 Dec 9;11(12):e0166439. doi: 10.1371/journal.pone.0166439. eCollection 2016. PMID 27936001
- [Background] Woods DL, Wyma JM, Herron TJ, Yund EW. A Computerized Test of Design Fluency. PLoS One. 2016 May 3;11(5):e0153952. doi: 10.1371/journal.pone.0153952. eCollection 2016. PMID 27138985
- [Background] Woods DL, Yund EW, Wyma JM, Ruff R, Herron TJ. Measuring executive function in control subjects and TBI patients with question completion time (QCT). Front Hum Neurosci. 2015 May 19;9:288. doi: 10.3389/fnhum.2015.00288. eCollection 2015. PMID 26042021